CLINICAL TRIAL: NCT05264181
Title: Long Term Outcomes Following Transcatheter Pulmonary Valve Implantation With SAPIEN 3 Valve : a Multicentre International Study
Brief Title: Transcatheter Pulmonary Valve Implantation With SAPIEN 3 Valve
Acronym: EUROPULMS3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Collaborators: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: 2022-564
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Valve; Failure; Percutaneous Pulmonary Valve Implantation; Infective Endocarditis; Congenital Heart Disease
Keywords: percutaneous pulmonary valve implantation; SAPIEN 3; transcatheter pulmonary valve replacement; infective endocarditis; Congenital Heart Disease
MeSH Terms: conditions — Endocarditis; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Percutaneous pulmonary valve implantation — Percutaneous pulmonary valve implantation using SAPIEN 3 valve in the context of routine care of patients with congenital heart diseases

SUMMARY:
Background Transcatheter pulmonary valve implantation (TPVI) is indicated to treat right ventricular outflow tract dysfunction in patients with congenital heart diseases. Long-term outcomes following this procedure using the new generation SAPIEN 3 valve is little known.

Purpose This study aims to report mid-term outcomes in a large cohort of patients who had TPVI using the SAPIEN 3 valve.

Methods We designed a retrospective multicentre observational registry of patients undergoing TPVI with the SAPIEN 3 valve across centres in Europe, Middle-east and Canada. Patient-related, procedural, and mid-term outcomes data will be characterized.

DETAILED DESCRIPTION:
1. INTRODUCTION Percutaneous pulmonary valve implantation (PPVI) is effective to treat right ventricle outflow (RVOT) dysfunction. First reported by Bonhoeffer et al. in 2000, PPVI extends the lifespan of an existing RVOT revision and delays the need for repeat surgical intervention. First limited to patients with dysfunctional right-ventricle to pulmonary artery conduit, its feasibility was extended to patients with bioprosthesis, small expandable conduits and native RVOT. In select patients, it is nowadays a first-line approach to PV replacement. With longer follow-up, some issues arose such as the incidence of infective endocarditis (IE). It remains highly debatable if the risk of IE varied according to the type of implanted valve. Tricuspid valve injuries were also reported while advancing a valve without covering along the right heart cavities. However, most of the current evidence has been gathered using the early generation Melody (Medtronic Inc., Minneapolis, MN) or Edwards SAPIEN valves (Edwards Lifesciences, Irvine, CA).

   Ongoing prosthesis improvement programmes have led to the availability of the SAPIEN 3 (S3), a bovine pericardial valve mounted on a fatigue-resistant cobalt chromium alloy stent with inclusion of an outer polyethylene terephthalate skirt, available in 20, 23, 26 and 29 mm in diameter. First implanted in 2014 in pulmonary position and subsequently described in preliminary multicentre reports, PPVI with the S3 valve appears to be safe and feasible in a wide range of patients with congenital heart defects, including those with large native RVOT. Use of this valve and its smooth deflectable Commander delivery system has been shown to facilitate PPVI, together with the use of a long introducer delivery sheath. The procedures resulted in good short-term haemodynamic and functional outcomes, with very few adverse events, paving the way for worldwide implantation of the S3 valve in the pulmonic position. Furthermore, while prestenting is systematically recommended before implanting a Melody valve to decrease the risk of stent fracture during follow-up, S3 design and radial strength resulted in a modification of implantation method with decreased prestenting indications. However, positive safety and efficacy outcomes remains to be demonstrated over the longer term. There is currently little formal data on S3 implantation in the pulmonic position over few months. The objective of the present multicentre registry analysis was to explore safety, feasibility, and haemodynamic outcomes of PPVI using the S3 to up to five years.
2. METHODS We designed a retrospective multicentre cohort study including all consecutives PPVI of a S3 valve between 2014 and decembre 2021 in European, Canadian and middle-east centres.

   The study was approved by an ethical committees (GERM IRB 00012157, reference 543, 27 October 2021) and performed in accordance with the Declaration of Helsinki and its amendments.

   2.1 Centres These centres are situated in Europe (France, United-Kingdom, Germany, Italy, Spain, Switzerland, Poland), the Middle East (Turkey, Israel), and Canada. No minimum requirements pertaining to number of implants or operator experience are specified.

   2.2 Patients Inclusion criteria were a clinical indication for PPVI and a prior implantation of the S3 in the pulmonic position, with the decision to perform the procedure taken independently. So as to represent the broadest possible spectrum of patients undergoing PPVI, no further inclusion/exclusion criteria were stipulated. PPVI is usually indicated in symptomatic patients or those with evidence of RV or left ventricular systolic dysfunction, severe RV enlargement with an indexed RV end-diastolic volume of greater than 160 mL/m2, or an indexed RV end-systolic volume of greater than 80 mL/m2 and those with decreases in exercise capacity.

   PPVI was performed using SAPIEN 3 valve in all cases. The SAPIEN 3 valve is characterized by a trileaflet valve crafted from bovine pericardium treated with the same ThermaFix process as Carpentier-Edwards surgical valves. The valve is sutured to a cobalt-chromium stent frame with optimized cell design to minimize profile and improve radial strength. Additionally, the SAPIEN 3 has an outer polyethylene terephthalate skirt which decreases the incidence of paravalvular leak. The SAPIEN 3 valve is available in 20- 23-, 26-, and 29-mm sizes and is introduced using the Commander delivery system (14 and 16-Fr expandable sheaths). It has obtained CE mark in 2021.

   2.3 Data collection Given the wide range of patients represented in the study, the Pulmonic S3 electronic case report form (eCRF) was designed to accommodate the broadest possible spectrum of clinical settings in which PPVI may be indicated. As such, the data collected reflects the site's standard procedures, including but not limited to physical assessments, ECGs, laboratory testing, and cardiac imaging. Data entry was performed by the treating physician or study nurse through retrospective appraisal of medical records.

   Data regarding patient demographics, underlying diagnoses and RVOT anatomies were collected for the period prior to PPVI, with peri-procedural details and outcomes also documented. Follow-up time points for the assessment of adverse events and functional outcomes were 30 days, six months, one and two years. Data were subjected to regular automatic and manual checks for plausibility and completeness.

   2.4 Outcomes and definitions Key haemodynamic and functional outcomes included changes in the peak systolic gradient over RVOT; degree of pulmonary regurgitation following PPVI. Feasibility was assessed according to procedural success (defined as successful implantation of a single valve at the intended location and retrieval of the delivery catheter), while safety outcomes included the rates of periprocedural technical complications (device malfunction [defined as failure to meet performance specifications or otherwise perform as expected]; valve dislocation requiring surgical intervention; and stent dislocation), periprocedural adverse events (significant bleeding; arrhythmia requiring pacing, drugs or cardioversion; conduit/RVOT rupture requiring emergency stenting or surgery; significant neurological impairment [based on clinical assessment; coronary compression; myocardial infarction; pulmonary embolism; and periprocedural death).

   2.5 Statistics Data are presented as descriptive data summaries. Categorical variables are expressed as absolute numbers and frequencies (%), while continuous variables are expressed as means with standard deviations (SD) and minimum-maximum data ranges.
3. RESULTS 3.1 Patient characteristics will be displayed 3.2 Procedural characteristics will be displayed 3.3 Periprocedural outcomes and safety will be reported

   * What is known:

Percutaneous pulmonary valve implantation is safe and effective to treat right ventricle outflow tract dysfunction in patients with congenital heart diseases A wide spectrum of devices are being used currently. The new-generation SAPIEN 3 valve has recently been labelled for percutaneous pulmonary valve implantation.

• What the Study will Add: SAPIEN 3 Three and Five-years freedom from secondary pulmonary valve replacement will be reported SAPIEN 3 Annualized Incidence of infective endocarditis will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patient with congenital heart disease, dysfunctional right ventricle outflow tract and indications for percutaneous pulmonary valve replacement as indicated by international guidelines-
* Patient having a valve replacement using a SAPIEN 3 valve

Exclusion Criteria:

* Patient having a valve replacement using a SAPIEN XT valve
* Patient having a valve replacement using a Melody valve
* Patient having a valve replacement using a Harmony valve
* Patient having a valve replacement using a Venus-P valve
* Patient refusing participation to the study

Ages: 5 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion criteria were a clinical indication for PPVI in the pulmonic position, with the decision to perform the procedure taken independently. So as to represent the broadest possible spectrum of patients undergoing PPVI, no further inclusion/exclusion criteria were stipulated. PPVI is usually indicated in symptomatic patients with congenital heart diseases or those with evidence of RV or left ventricular systolic dysfunction, severe RV enlargement with an indexed RV end-diastolic volume of greater than 160 mL/m2, or an indexed RV end-systolic volume of greater than 80 mL/m2 and those with decreases in exercise capacity.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
secondary pulmonary valve replacement | 5 years
  annualized incidence of secondary valve replacement by catheterization or surgery for SAPIEN 3 valve failure

SECONDARY OUTCOMES:
Infective endocarditis | 5 years
  Annualized incidence of infective endocarditis on the SAPIEN 3 Vave
Thrombosis | 5 years
  Annualized incidence of pulmonary vavle thrombosis following PPVI with Sapien 3 valve

CONTACTS AND LOCATIONS:
Overall Officials: Alain Fraisse, MD, PhD, Study Director — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No